CLINICAL TRIAL: NCT02554162
Title: Chewy Satiety - the Interplay Between Food Structure, Oral Processing and Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VTT Technical Research Centre of Finland (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Chewy
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2015-12

CONDITIONS: Subjective Appetite and Satiety
Keywords: Satiety, appetite, wholegrain rye

STUDY DESIGN:
Who Masked: Participant

ARMS (5):
- Extruded wholegrain rye flakes (Active Comparator): Rye products with varying structures
  Interventions: Other: Rye products with varying structures
- Extruded wholegrain rye puffs (Active Comparator): Rye products with varying structures
  Interventions: Other: Rye products with varying structures
- Fresh wholegrain rye bread (Active Comparator): Rye products with varying structures
  Interventions: Other: Rye products with varying structures
- Wholegrain rye beverage (Active Comparator): Rye products with varying structures
  Interventions: Other: Rye products with varying structures
- Fresh wheat bread (Active Comparator): Rye products with varying structures
  Interventions: Other: Rye products with varying structures

INTERVENTIONS:
Other: Rye products with varying structures — The satiating effect of rye products with various structures will be studied

SUMMARY:
This study examines if there are differences in satiety responses between structurally different wholegrain rye products.

DETAILED DESCRIPTION:
The study consists of a satiety trial and mastication trial. The satiety trial consists of five study visits. Five cereal products with berry soup are presented in random order for each subject serving one of them in each study visit (crossover study design). Each meal consists of rye product or wheat bread providing 190 kcal of energy and of 3 dl berry soup (3 dl) providing 140 kcal of energy. The participants are instructed to evaluate their satiety and related sensations before eating the test food, right after eating and then every 30 min until 210 min after breakfast consumption. The evaluated sensations are hunger, fullness, satiety, desire to eat and prospective food consumption ("How much would you be able to eat right now?"), "thirstiness", "mood", "vigourosness" and "pleasantness"."Pleasantness" will be evaluated only right after eating the test food.

Cereal food samples with 3-digit number codes will be offered to each participant in a random order in mastication trial. The study products are rye products with varying structures. First the participant is asked to evaluate the expected satiety of the product (How filling would you expect this portion to be on a scale from 0 (=not full at all) to 10 (=extremely full)). Secondly the same food will be served to the participant in three portions and the participant will be asked to masticate each portion until she considers it to be ready for swallowing. Instead of swallowing the bolus will be expectorated to a plastic container which is kept on ice. The mastication process is characterized by measuring electrical activity of facial muscles by electromyography (EMG). The mastication process will be video-recorded to support data handling.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-25 kg/m2
* Habit of eating breakfast

Exclusion Criteria:

* Significant changes in body weight (+ or - 4 kg) during the previous year
* Smoking
* Pregnant or lactating
* Missing teeth (except 3rd molars)
* Acute temporomandibular disorders (TMD)
* Dietary restrictions possibly affecting the study (celiac disease, allergies or aversions to cereal foods/high carbohydrate foods)
* Abnormal eating behaviour (according to EDDS (Eating Disorder Diagnostic Scale))

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Postprandial satiety, assessed using 10 cm visual analogue scale (0=not at all, 10=Extremely) | In every 30 min until 210 min after consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Aalto University, Espoo, Finland